CLINICAL TRIAL: NCT00612417
Title: A Randomised, Double-blind and Placebo-controlled Study Investigating the Pharmacodynamic Effects of Administration of Recombinant Human Factor VIII in Healthy Male Subjects Treated With the Monoclonal Anti-factor VIII Antibody, TB-402
Brief Title: Effect of Recombinant FVIII in Healthy Male Subjects Treated With TB-402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Collaborators: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TB-402-002
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Interaction with recombinant FVIII
MeSH Terms: interventions — TB 402

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): recombinant FVIII
  Interventions: Drug: Administration of recombinant FVIII/placebo in healthy male subjects treated with TB-402
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Administration of recombinant FVIII/placebo in healthy male subjects treated with TB-402

INTERVENTIONS:
Drug: Administration of recombinant FVIII/placebo in healthy male subjects treated with TB-402 — Administration of recombinant FVIII/placebo in healthy male subjects treated with TB-402

SUMMARY:
Single administration of recombinant FVIII/placebo in healthy male subjects who have been treated with a single dose of anti-factor VIII antibody, TB-402

ELIGIBILITY:
Inclusion Criteria include:

* Males 18 to 45 years of age
* Healthy according to medical history, physical exam, ECG, blood pressure and heart rate, and laboratory profile of blood and urine

Exclusion Criteria include:

* Self or family history of cardiovascular or pulmonary disorder, or coagulation or bleeding disorders or reasonable suspicion of vascular malformations e.g. cerebral haemorrhage, aneurysm or premature stroke
* History of important bleeding episodes
* Previous allergic reaction to immunoglobulin
* Present or previous history of severe allergy, for example asthma or anaphylactic reactions
* FVIII:C <50% or >150% at screening
* Clinically significant out of range values for any coagulation test during screening
* Received prescribed medication, over the counter medication or herbal medicines within 14 days of receipt of TB-402

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Changes in coagulation parameters after rFVIII administration | To study end

SECONDARY OUTCOMES:
PD of TB-402, safety of TB-402 alone and with rFVIII, PK of FVIII in rFVIII-treated subjects, changes in coagulation parameters after TB-402 administration | To study end

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Jensen, MD, PhD, Principal Investigator — Cyncron CRU
Locations (1):
- Cyncron CRU, Copenhagen, Denmark